CLINICAL TRIAL: NCT00056303
Title: Specialized Mental Health Services for Foster Infants
Brief Title: Mental Health Services for Foster and Adopted Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Dozier, UNIDEL-Amy E dupont Professor, Psychology, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01MH052135 (NIH); R01MH052135 (NIH); DSIR 84-CTCT
Record Dates: First submitted 2003-03-10; First posted 2003-03-11 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Problem Behaviors; Attention Deficit Hyperactivity Disorder; Depression
Keywords: Attachment; Intervention; Prevention
MeSH Terms: conditions — Problem Behavior; Attention Deficit Disorder with Hyperactivity; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attachment and Biobehavioral Catch-up (Experimental): Attachment and Biobehavioral Catch-up targets nurturance, synchrony, and non-frightening behavior, as well as providing caregivers with help calming toddlers.
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up
- Developmental Education for Families (Active Comparator): Developmental Education for Families targets providing cognitive stimulation to their children.
  Interventions: Behavioral: Developmental Education for Families

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up — Attachment and Biobehavioral Catch-up is a 10 session in-home intervention that targets synchrony, nurturance, and calming parental behavior.
  Arms: Attachment and Biobehavioral Catch-up
Behavioral: Developmental Education for Families — Developmental Education for Families is a 10-session in home intervention that targets children's cognitive development.
  Arms: Developmental Education for Families

SUMMARY:
This study will determine the effectiveness of a relationship-based intervention in improving the interaction between caregivers and young children placed in their care.

DETAILED DESCRIPTION:
Infants and toddlers who are placed into foster or adoptive care often exhibit a number of behavioral, emotional, and physiological problems. In the absence of specialized services, problems in the relationship between caregiver and child may develop; problems in the child's functioning often persist and are exacerbated. This study will attempt to alleviate the attachment and regulatory difficulties that affect many young children placed into care.

Children are randomly assigned to either an experimental group or to a treatment control group for 3 years. The experimental group focuses on relational issues; the control group focuses on cognitive development. Caregivers receiving the relational intervention are trained to provide nurturing care, and to help children learn to develop adequate regulatory skills. Caregivers in the treatment control group receive training designed to enhance children's cognitive development. Caregivers in both groups will receive 10 home visits. Observations of children and parents are used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* Toddler placed into foster care
* Resident of Delaware and surrounding counties in Pennsylvania and Maryland

Exclusion Criteria:

* Significant medical problems

Ages: 20 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2002-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Attachment | Annually
  The Preschool Strange Situation is conducted annually.

SECONDARY OUTCOMES:
Executive Functioning | Annually
  Disruptive Behaviors-Diagnostic Observation Schedule (DB-DOS) is used to assess problem behaviors. The DB-DOS consists of a series of challenging tasks that ask the child to inhibit prepotent behaviors and regulate emotions.
Diurnal production of cortisol | Annually
  Three days of saliva sampling at wake-up and bedtime.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dozier, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No